CLINICAL TRIAL: NCT02965534
Title: Evaluation of a Night Spectacle Correction Concerning an Improvement of Mesopic Vision Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Applied Sciences Jena (Other)
Collaborators: IGA OPTIC EG (Unknown)
Responsible Party: Principal Investigator, Stephan Degle, Prof. Dr., University of Applied Sciences Jena
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IGAMYO
Record Dates: First submitted 2016-11-14; First posted 2016-11-16 (Estimated); Results first posted 2019-02-28 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2018-10

CONDITIONS: Myopia-Night Blindness
Keywords: night vision; mesopic visual acuity; aberrometry; mesopic spectacle correction; night myopia
MeSH Terms: conditions — Night blindness, congenital stationary | interventions — Eyeglasses

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Night Spectacle Correction (Experimental): Refraction for this glasses was obtained at low luminance.
  Interventions: Device: Spectacle/Glasses
- Spectacle Correction for photopic light conditions (Active Comparator): Refraction for this glasses was obtained at high luminance level.
  Interventions: Device: Spectacle/Glasses

INTERVENTIONS:
Device: Spectacle/Glasses

SUMMARY:
Reduced quality of vision and glare in twilight or night are frequently mentioned complaints within the optometric examination. A reason for these problems could be a myopic refractive shift in dark light conditions, commonly known as night myopia or twilight myopia.

The aim of this study was to investigate whether quality of vision in twilight or night could be improved by a spectacle correction optimized for mesopic light conditions. Moreover, objective refraction in large pupils measured by aberrometry was compared to subjective mesopic refraction.

DETAILED DESCRIPTION:
After obtaining informed consent, aberrometry was performed in a darkened room (0.1 lux). Subjective photopic refraction and visual acuity were measured before light was turned off and mesopic refraction was obtained after a dark adaptation period of five minutes. Finally, frames and lenses were fitted by a centration system. Lens grinding was executed centralized by a grinding workshop. In the course of this study, subjects were randomly assigned to wear two glasses double-masked in turn. One with photopic subjective refraction data and another with mesopic subjective refraction data. Both were worn for 14 ± 2 days each.

Follow Up 1:

After two weeks, participants were asked for their subjective experiences with the first correction by a visual analogue scale questionnaire. After the evaluation, glasses were changed.

Follow Up 2:

Two weeks later, subjective experiences were evaluated again. After visual analogue scale questionnaire, subjects were asked to compare the two glasses concerning quality of mesopic vision and subjective safety level during night driving.

ELIGIBILITY:
Inclusion Criteria:

* Visual Acuity at least 0.8 (5/6)
* Binocular Vision

Exclusion Criteria:

* refraction more than sph +/- 6 D and cyl 2 D
* Difference between habitual correction and actual refraction more than 0.5 D
* Medication with an influence on visual system
* Disease or eye disease with an effect on the visual system
* pregnancy or other hormonal variances
* influence of drugs
* mental handicap

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-10; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Degle, Prof., Principal Investigator — University of Applied Sciences Jena
Locations (3):
- Germany (3):
  - Degle Optometry, Augsburg, Bavaria
  - Hessler Optometry, Klingenberg am Main, Bavaria
  - University of Applied Sciences, Jena, Thuringia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Night Spectacle Correction - Photopic Spectacle Correction: This arm has tested first the mesopic spectacle correction for 2 weeks and after this time the ("standard") photopic spectacle correction for two weeks
  Cross Over Design!
- Photopic Spectacle Correction - Night Spectacle Correction: This arm has tested first the standard photopic spectacle correction for two weeks and after this time the mesopic spectacle correction for two weeks
  Cross Over Design!
Period: Overall Study
Arm/Group | Night Spectacle Correction - Photopic Spectacle Correction | Photopic Spectacle Correction - Night Spectacle Correction
Started | 45 (test period: 14 days with each test glasses) | 55 (test period: 14 days with each test glasses)
Completed | 45 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: All subjects were included in Baseline and all investigations were obtained at these 100 subjects
Arm/Group | All Subjects
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78
  Male | 22
Aberrometry Spherical Equivalent (SE) small pupil OD [Mean (Standard Deviation); unit: D] — OD = right eye. Spherical Equivalent was calculated with data of an aberrometer (VISIONIX VX120 family).
  Spherical Equivalent is calculated by (sph + 0.5*cyl).
  D | -1.44 (1.74)
Aberrometry SE at small pupil OS [Mean (Standard Deviation); unit: D] — SE = Spherical Equivalent. OS = left eye. Spherical Equivalent was calculated with data of an aberrometer (VISIONIX VX120 family).
  Spherical Equivalent is calculated by (sph + 0.5*cyl).
  D | -1.36 (1.86)
Subjective photopic Refraction SE OD [Mean (Standard Deviation); unit: D] — SE = Spherical Equivalent OD = Right Eye
  Subjective Refraction measured in a photopic luminance level (comparable to an eye examination for new glasses). Spherical Equivalent was calculated with data of subjective refraction.
  Spherical Equivalent is calculated by (sph + 0.5*cyl).
  D | -1.10 (1.69)
Subjective photopic Refraction SE OS [Mean (Standard Deviation); unit: D] — SE = Spherical Equivalent OS = Left Eye
  Subjective Refraction measured in a photopic luminance level (comparable to an eye examination for new glasses). Subjective Refraction measured in a photopic luminance level. Spherical Equivalent was calculated with data of subjective refraction.
  Spherical Equivalent is calculated by (sph + 0.5*cyl).
  D | -1.03 (1.79)
Photopic Visual Acuity OD [Median (Full Range); unit: logMAR Visual Acuity] — Best Corrected Visual Acuity in a photopic luminance. OD = Right Eye
  0.0 corresponds to a Snellen Visual Acuity 20/20, 0.1 to 20/25, 0.2 to 20/32,
  -0.1 to 20/16, etc.
  logMAR Visual Acuity | -0.1 [-0.2 to 0.1]
Photopic Visual Acuity OS [Median (Full Range); unit: logMAR Visual Acuity] — Best Corrected Visual Acuity in a photopic luminance OS = Left Eye. 0.0 corresponds to a Snellen Visual Acuity 20/20, 0.1 to 20/25, 0.2 to 20/32,
  -0.1 to 20/16, etc
  logMAR Visual Acuity | -0.1 [-0.2 to 0.1]
Binocular photopic Visual Acuity [Median (Full Range); unit: logMAR Visual Acuity] — Best Corrected Visual Acuity in a photopic luminance, binocular. 0.0 corresponds to a Snellen Visual Acuity 20/20, 0.1 to 20/25, 0.2 to 20/32,
  -0.1 to 20/16, etc.
  logMAR Visual Acuity | -0.2 [-0.3 to 0]
Mesopic Visual Acuity with photopic refraction OD [Median (Full Range); unit: logMAR Visual Acuity] — Visual Acuity measured in a mesopic luminance, wearing refraction values measured in photopic luminance OD = Right Eye. 0.0 corresponds to a Snellen Visual Acuity 20/20, 0.1 to 20/25, 0.2 to 20/32,
  -0.1 to 20/16, etc.
  logMAR Visual Acuity | 0.1 [0 to 0.3]
Mesopic Visual Acuity with photopic refraction OS [Median (Full Range); unit: logMAR Visual Acuity] — Visual Acuity measured in a mesopic luminance, wearing refraction values measured in photopic luminance OS = Left Eye. 0.0 corresponds to a Snellen Visual Acuity 20/20, 0.1 to 20/25, 0.2 to 20/32,
  -0.1 to 20/16, etc.
  logMAR Visual Acuity | 0.1 [-0.1 to 0.4]
Mesopic Visual Acuity with photopic refraction Binocular [Median (Full Range); unit: logMAR Visual Acuity] — Visual Acuity measured in a mesopic luminance, wearing refraction values measured in photopic luminance Binocular.
  0.0 corresponds to a Snellen Visual Acuity 20/20, 0.1 to 20/25, 0.2 to 20/32,
  -0.1 to 20/16, etc.
  logMAR Visual Acuity | 0.1 [-0.1 to 0.3]
Subjective Mesopic Refraction SE OD [Mean (Standard Deviation); unit: D] — Mesopic Refraction measured in mesopic luminance (comparable to an eye examination for new glasses in a darkened room).
  OD = Right Eye SE = Spherical Equivalent
  D | -1.42 (1.69)
Subjective Mesopic Refraction SE OS [Mean (Standard Deviation); unit: D] — Mesopic Refraction measured in mesopic luminance (comparable to an eye examination for new glasses in a darkened room).
  OS = Right Eye SE = Spherical Equivalent
  D | -1.37 (1.76)
Mesopic Visual Acuity with Mesopic Refraction OD [Median (Full Range); unit: logMAR Visual Acuity] — Best corrected visual acuity after refraction in mesopic luminance OD = Right Eye. 0.0 corresponds to a Snellen Visual Acuity 20/20, 0.1 to 20/25, 0.2 to 20/32,
  -0.1 to 20/16, etc.
  logMAR Visual Acuity | 0.0 [-0.1 to 0.2]
Mesopic Visual Acuity with Mesopic Refraction OS [Median (Full Range); unit: logMAR Visual Acuity] — Best corrected visual acuity after refraction in mesopic luminance OS = Left Eye. 0.0 corresponds to a Snellen Visual Acuity 20/20, 0.1 to 20/25, 0.2 to 20/32,
  -0.1 to 20/16, etc.
  logMAR Visual Acuity | 0.0 [-0.1 to 0.2]
Mesopic Visual Acuity with Mesopic Refraction Binocular [Median (Full Range); unit: logMAR Visual Acuity] — Best corrected visual acuity after refraction in mesopic luminance Binocular. 0.0 corresponds to a Snellen Visual Acuity 20/20, 0.1 to 20/25, 0.2 to 20/32,
  -0.1 to 20/16, etc.
  logMAR Visual Acuity | 0.0 [-0.2 to 0.2]
Spherical Aberration OD [Mean (Standard Deviation); unit: µm] — Measured by Aberrometry OD = Right Eye
  µm | 0.100 (0.15)
Spherical Aberration OS [Mean (Standard Deviation); unit: µm] — Measured by Aberrometry OS = Left Eye
  µm | 0.093 (0.14)
Max. pupil size aberrometry OD [Mean (Standard Deviation); unit: mm] — measured by aberrometry OD = Right Eye
  mm | 5.6 (0.7)
Max. pupil size aberrometry OS [Mean (Standard Deviation); unit: mm] — measured by aberrometry OS = Left Eye
  mm | 5.8 (0.8)
Aberrometry Spherical Equivalent (SE) large pupil OD [Mean (Standard Deviation); unit: D] — OD = Right Eye. Spherical Equivalent was calculated with data of an aberrometer (VISIONIX VX120 family).
  Spherical Equivalent is calculated by (sph + 0.5*cyl). SE value of max. pupil size.
  D | -1.67 (1.68)
Aberrometry Spherical Equivalent (SE) large pupil OS [Mean (Standard Deviation); unit: D] — OS = Left Eye. Spherical Equivalent was calculated with data of an aberrometer (VISIONIX VX120 family).
  Spherical Equivalent is calculated by (sph + 0.5*cyl). SE value of max. pupil size.
  D | -1.58 (1.83)
Pupil size in photopic light conditions OD [Mean (Standard Deviation); unit: mm] — Measured by Infra Red Camera in photopic conditions OD = Right Eye
  mm | 4.3 (1.0)
Pupil size in photopic light conditions OS [Mean (Standard Deviation); unit: mm] — Measured by Infra Red Camera in photooic conditions. OS = Left Eye
  mm | 4.3 (1.0)
Pupil size in mesopic light conditions OD [Mean (Standard Deviation); unit: mm] — Measured by Infra Red Camera in mesopic conditions. OD = Right Eye
  mm | 6.5 (1.4)
Pupil size in mesopic light conditions OS [Mean (Standard Deviation); unit: mm] — Measured by Infra Red Camera in mesopic conditions OS = Left Eye
  mm | 6.6 (1.4)
J0 Aberrometry OD small pupil [Mean (Standard Deviation); unit: D] — J0 = Astigmatism component OD = Right Eye
  D | -0.03 (0.26)
J0 Aberrometry OS small pupil [Mean (Standard Deviation); unit: D] — J0 = Astigmatism component OS = Left Eye
  D | 0.01 (0.29)
J45 Aberrometry OD small pupil [Mean (Standard Deviation); unit: D] — J45 = Astigmatism component OD = Right Eye
  D | 0.01 (0.35)
J45 Aberrometry OS small pupil [Mean (Standard Deviation); unit: D] — J45 = Astigmatism component OS = Left Eye
  D | 0.01 (0.30)
J0 Aberrometry OD large pupil [Mean (Standard Deviation); unit: D] — J0 = Astigmatism component OD = Right Eye
  D | -0.02 (0.31)
J0 Aberrometry OS large pupil [Mean (Standard Deviation); unit: D] — J0 = Astigmatism component OS = Left Eye
  D | 0.03 (0.31)
J45 Aberrometry OD large pupil [Mean (Standard Deviation); unit: D] — J45 = Astigmatism component OD = Right Eye
  D | 0.01 (0.31)
J45 Aberrometry OS large pupil [Mean (Standard Deviation); unit: D] — J45 = Astigmatism component OS = Left Eye
  D | 0.01 (0.30)
J0 Subjective Photopic Refraction OD [Mean (Standard Deviation); unit: D] — J0 = Astigmatism component Calculated after performing cross-cylinder method OD = Right Eye
  D | -0.01 (0.26)
J0 Subjective Photopic Refraction OS [Mean (Standard Deviation); unit: D] — J0 = Astigmatism component Calculated after performing cross-cylinder method OS = Left Eye
  D | 0.03 (0.23)
J45 Subjective Photopic Refraction OD [Mean (Standard Deviation); unit: D] — J45 = Astigmatism component Calculated after performing cross-cylinder method OD = Right Eye
  D | 0.01 (0.21)
J45 Subjective Photopic Refraction OS [Mean (Standard Deviation); unit: D] — J45 = Astigmatism component Calculated after performing cross-cylinder method OS = Left Eye
  D | 0.05 (0.23)
J0 Subjective Mesopic Refraction OD [Mean (Standard Deviation); unit: D] — J0 = Astigmatism component Calculated after performing cross-cylinder method in a darkened room OD = Right Eye
  D | -0.01 (0.25)
J0 Subjective Mesopic Refraction OS [Mean (Standard Deviation); unit: D] — J0 = Astigmatism component Calculated after performing cross-cylinder method in a darkened room OS = Left Eye
  D | 0.03 (0.27)
J45 Subjective Mesopic Refraction OD [Mean (Standard Deviation); unit: D] — J45 = Astigmatism component Calculated after performing cross-cylinder method in a darkened room OD = Right Eye
  D | -0.02 (0.25)
J45 Subjective Mesopic Refraction OS [Mean (Standard Deviation); unit: D] — J45 = Astigmatism component Calculated after performing cross-cylinder method in a darkened room OS = Left Eye
  D | -0.01 (0.22)

OUTCOME MEASURES:

1. Primary Outcome: Night Myopia
Description: Value of refractive shift (SE) when changing luminance from a photopic to a mesopic level.
  At Baseline, participants were not separated into arms as the Randomization Process was carried out at a later time point after participants picked up study glasses. Therefore, data are presented for All Participants in one Arm/Group.
Time Frame: Baseline only
Measure: Mean (Standard Deviation); unit: D
Arm/Group | All Subjects
Number analyzed (Participants) | 100
D
  Right Eye (OD): shift in SE | -0.30 (0.2)
  Left Eye (OS): shift in SE | -0.32 (0.21)

2. Secondary Outcome: Mesopic Visual Acuity Improvement
Description: Difference of visual acuity (monocular and binocular) in a darkened room (0.1 lux) after a dark adaption period of 5 min. with photopic spectacle correction ("classic" refraction obtained in photopic light conditions) compared to mesopic spectacle correction (correction of night myopia)
  Scale: logMAR visual acuity, using Landolt C optotypes.
  At Baseline, participants were not separated into arms as the Randomization Process was carried out at a later time point after participants picked up study glasses. Therefore, data are presented for All Participants in one Arm/Group.
Time Frame: Baseline only
Measure: Median (Full Range); unit: logMAR visual acuity
Arm/Group | All Subjects
Number analyzed (Participants) | 100
logMAR visual acuity
  Right Eye (OD): visual acuity improvement | 0.1 [0 to 0.4]
  Left Eye (OS): visual acuity improvement | 0.1 [0 to 0.3]
  Binocular visual acuity improvement | 0.1 [0 to 0.3]

3. Secondary Outcome: Subjective Vision Comfort in Dark Light Conditions
Description: Evaluation of subjective perceived vision comfort with the study and control glasses.
  Both glasses (study and control glasses) were tested for two weeks each. After the two weeks test, each of the glasses was evaluated. For evaluation a visual analogue scale questionnaire (Scale 0 - 100) was used.
  Question:
  How would you evaluate vision comfort with the tested glasses in dark light conditions? Answer: visual analogue scale slider from 0 (insufficient) to 100 (very good)
Time Frame: Test Period (4 weeks)
Measure: Mean (Standard Deviation); unit: scores on a scale (0 to 100)
Groups:
- Night Spectacle Correction: Refraction for this glasses was obtained at low luminance.
  Spectacle/Glasses
- Spectacle Correction for Photopic Light Conditions: Refraction for this glasses was obtained at high luminance level.
  Spectacle/Glasses
Arm/Group | Night Spectacle Correction | Spectacle Correction for Photopic Light Conditions
Number analyzed (Participants) | 100 | 100
scores on a scale (0 to 100) | 60 (31) | 73 (26)

4. Secondary Outcome: Subjective Vision Sharpness in Dark Light Conditions
Description: Evaluation of subjective perceived vision sharpness with the study and control glasses.
  Both glasses (study and control glasses) were tested for two weeks each. After the two weeks test, each of the glasses was evaluated. For evaluation a visual analogue scale questionnaire (Scale 0 - 100) was used.
  Question:
  How would you evaluate vision sharpness with the tested glasses in dark light conditions? Answer: visual analogue scale slider from 0 (insufficient) to 100 (very good)
Time Frame: Test Period (4 weeks)
Measure: Mean (Standard Deviation); unit: evaluation points (0 to 100)
Arm/Group | Night Spectacle Correction | Spectacle Correction for Photopic Light Conditions
Number analyzed (Participants) | 100 | 100
evaluation points (0 to 100) | 59 (30) | 73 (27)

5. Secondary Outcome: Subjective Glare Sensitivity in Dark Light Conditions
Description: Evaluation of subjective perceived glare sensitivity with the study and control glasses.
  Both glasses (study and control glasses) were tested for two weeks each. After the two weeks test, each of the glasses was evaluated. For evaluation a visual analogue scale questionnaire (Scale 0 - 100) was used.
  Question:
  How would you evaluate glare sensitivity with the tested glasses in dark light conditions? Answer: visual analogue scale slider from 0 (no glare) to 100 (strong glare)
Time Frame: Test Period (4 weeks)
Measure: Mean (Standard Deviation); unit: scores on a scale (0 to 100)
Arm/Group | Night Spectacle Correction | Spectacle Correction for Photopic Light Conditions
Number analyzed (Participants) | 100 | 100
scores on a scale (0 to 100) | 48 (32) | 37 (31)

6. Secondary Outcome: Subjective Driving Safety in Dark Light Conditions
Description: Evaluation of subjective perceived driving safety sense with the study and control glasses.
  Both glasses (study and control glasses) were tested for two weeks each. After the two weeks test, each of the glasses was evaluated. For evaluation a visual analogue scale questionnaire (Scale 0 - 100) was used.
  Question:
  How would you evaluate driving safety sense when driving in twilight or night with the tested glasses? Answer: visual analogue scale slider from 0 (not safe) to 100 (very safe)
Time Frame: Test Period (4 weeks)
Measure: Mean (Standard Deviation); unit: scores on a scale (0 to 100)
Arm/Group | Night Spectacle Correction | Spectacle Correction for Photopic Light Conditions
Number analyzed (Participants) | 100 | 100
scores on a scale (0 to 100) | 57 (32) | 73 (25)

ADVERSE EVENTS:
Time Frame: study time
Arm/Group | Night Spectacle Correction | Spectacle Correction for Photopic Light Conditions
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No